CLINICAL TRIAL: NCT00360425
Title: A Phase 1 Active- and Placebo-Controlled Study of the Electrocardiogram Effects and Pharmacokinetics of Ferumoxytol in Healthy Men and Women
Brief Title: A Study of the Electrocardiogram Effects and Pharmacokinetics of Ferumoxytol in Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 62,745-9
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Anemia
Keywords: anemia; intravenous iron; pharmacokinetics; QTc
MeSH Terms: conditions — Anemia | interventions — Ferrosoferric Oxide; Moxifloxacin

INTERVENTIONS:
Drug: ferumoxytol
Drug: moxifloxacin
Drug: placebo

SUMMARY:
This study will define the effects of ferumoxytol on electrocardiogram (ECG) data as well as evaluate pharmacokinetics

DETAILED DESCRIPTION:
This trial will be conducted in order to provide an evaluation of the potential of ferumoxytol to cause cardiac arrhythmia in accordance with the International Conference on Harmonization (ICH) E14 guidance. The purpose of this trial is to define the effects of ferumoxytol on electrocardiogram (ECG) data. Pharmacokinetics will also be evaluated at multiple time points as specified. Subject safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females, 18 - 45 years of age, inclusive.
* Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum pregnancy test prior to enrollment into the trial.
* Subjects must give written informed consent and sign Health Insurance Portability and Accountability Act (HIPAA) guidelines to be in the study.
* Hemoglobin ≥ 10 g/dL and ≤ 16 g/dL for males and ≥ 10 g/dL and ≤ 14 g/dL for females.
* Transferrin saturation (TSAT) ≤ 35%
* Serum ferritin ≤ 100 ng/mL.
* Subjects must have a body mass index (BMI) between 19.0 and 30.0 kg/m2
* Subjects must have no clinically significant abnormal findings on the physical examination.

Exclusion Criteria:

* Subjects currently participating in a clinical trial with another investigational new drug or device or who have received an investigational new drug or device within 30 days or 5 half-lives (whichever is longer) prior to randomization into this study.
* Subjects who have been on parenteral or oral iron therapy within 30 days prior to dosing.
* Subjects with active infections requiring ongoing treatment.
* Subjects with a positive human immunodeficiency virus type 1 or type 2 (HIV-1 or HIV-2) antibody, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test.
* Abnormal liver function tests.
* Subjects who have had malignancy (except for non-melanoma of the skin), unless the subject has received curative treatment and has been disease free for > 2 years.
* Subjects with a history of risk factors for Torsades de pointes (TdP) [e.g., family history (parents or siblings) of long QT syndrome], history of fainting, unexplained loss of consciousness or convulsions.
* Clinically relevant abnormality on screening ECG
* Subjects who have a sustained supine systolic blood pressure (SBP) > 150 mmHg or < 90 mmHg or a diastolic blood pressure (DBP) < 45 or > 95 mmHg at screening or baseline.
* Subjects who have a pulse rate at rest of < 45 bpm or > 100 bpm.
* Subjects who are unable to stop smoking during the study (Day -1 to Day 7). Subjects who smoke 10 or more cigarettes a day.
* Excessive consumption (> 6 units per day) of food or beverages with xanthine or caffeine bases (e.g., tea, coffee, chocolate, cola; 1 unit of caffeine is contained in 6 oz of coffee, 4 oz of energy drink, 24 oz of cola, 12 oz of tea and 3 oz chocolate).
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men.
* Subjects with any allergies to iron products, moxifloxacin or multiple drug (two or more) allergies as reported by the subject or as determined by the investigator.
* Subjects who have taken medications [with the exception of Tylenol (acetaminophen) ≤ 2g/day, multi-vitamin that does not contain iron, hormonal contraception for females and hormone replacement therapy (HRT) in the case of menopausal subjects] within 7 days or 5 half-lives (whichever is longer) prior to randomization into this study.
* Subjects who the Investigator determines to have a medical status that would preclude the patient's participation in this protocol or who, for any reason, are deemed by the Investigator to be inappropriate for this study, including subjects who are unable to communicate or to cooperate during the study.
* Subjects with screening lab results that fall outside of the normal range limits and are considered to be clinically significant upon review by the Investigator.
* Subjects who have any condition possibly affecting drug absorption, [e.g., previous surgery on the gastrointestinal tract (including removal of parts of stomach, bowel, liver, gall bladder, or pancreas)].
* Subjects who have evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to these criteria (e.g., stable, mild joint disease) may be made following discussions with the Medical Monitor.
* Subjects who have donated blood or blood components within four weeks prior to the study. The Investigator should instruct subjects who participate in this study not to donate blood or blood components for four weeks after the completion of the study.
* Illegal drug users or subjects who have a history of drug abuse within the last 2 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174
Dates: Start 2006-05; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To define the effect of two doses of 510 mg ferumoxytol administered within 24 hours on the QTcI interval compared to placebo and to a single dose of 400 mg moxifloxacin.
To define the effect of two doses of 510 mg ferumoxytol administered within 24 hours on QT, QTcB, QTcF and heart rate (HR).
To assess the pharmacokinetics of two doses of 510 mg ferumoxytol administered within 24 hours.

SECONDARY OUTCOMES:
To describe the relationship between exposure to ferumoxytol and ECG parameters (QTcI, QT, QTcB, QTcF and HR).
To assess the safety and tolerability of a supratherapeutic dose of ferumoxytol (2 doses of 510 mg ferumoxytol administered within 24 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- [Background] Landry R, Jacobs PM, Davis R, Shenouda M, Bolton WK. Pharmacokinetic study of ferumoxytol: a new iron replacement therapy in normal subjects and hemodialysis patients. Am J Nephrol. 2005 Jul-Aug;25(4):400-10. doi: 10.1159/000087212. Epub 2005 Jul 28. PMID 16088081
- See also: National Kidney Foundation — http://www.kidney.org
- See also: National Anemia Action Council — http://www.anemia.org
- See also: Kidney Disease Outcomes Quality Initiative — http://www.kidney.org/Professionals/kdoqi/